CLINICAL TRIAL: NCT03525782
Title: A Clinical Study of Anti-MUC1 CAR T Cells and PD-1 Knockout Engineered T Cells for Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Anti-MUC1 CAR T Cells and PD-1 Knockout Engineered T Cells for NSCLC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangdong Pharmaceutical University (Other)
Collaborators: Guangzhou Anjie Biomedical Technology Co., Ltd. (Industry); University of Technology, Sydney (Other)
Responsible Party: Principal Investigator, Size Chen, Professor, The First Affiliated Hospital of Guangdong Pharmaceutical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-006
Record Dates: First submitted 2018-04-26; First posted 2018-05-16 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Lung Neoplasm Malignant; Non-small Cell Lung Cancer
Keywords: CAR-T cell therapy; MUC+; PD-1 Knockout; Non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Immunotherapy, Adoptive; pembrolizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- CAR-T (Experimental): Anti-MUC1 CAR-T cells will be prepared ex vivo and infused back to the patients.
  Interventions: Biological: CAR-T Cells
- CAR-T combining PD-1 knockout (Experimental): Anti-MUC1 CAR-T cells and PD-1 knockout Engineered T cells will be prepared ex vivo and infused back to the patients.
  Interventions: Biological: CAR-T Cells; Combination Product: CAR-T combining PD-1 Knockout; Biological: PD-1 knockout
- PD-1 knockout (Experimental): PD-1 knockout Engineered T cells will be prepared ex vivo and infused back to the patients.
  Interventions: Biological: PD-1 knockout
- PD-1 mAb (Active Comparator): Patients will be treated with a FDA approved monoclonal antibody for an identical course of treatment. This group will serve as PD-1 antibody treated group.
  Interventions: Drug: PD-1 mAb
- Sham Control (Placebo Comparator): Patient's T cells will be separate without genetic or engineered modification ex vivo and infused back to the patients.
  Interventions: Other: Sham control

INTERVENTIONS:
Biological: CAR-T Cells — Using the T cells from the patients to produce anti-MUC1 CAR-T Cells and then the cells will be infused back to the patients.
  Arms: CAR-T; CAR-T combining PD-1 knockout
Combination Product: CAR-T combining PD-1 Knockout — Using the T cells from the patients to prepare anti-MUC1 CAR-T Cells and PD-1 knockout T cells, then the cells will be infused back to the patients
  Arms: CAR-T combining PD-1 knockout
Biological: PD-1 knockout — Using the T cells from the patients to prepare PD-1 knockout T cells, then the cells will be infused back to the patients
  Arms: CAR-T combining PD-1 knockout; PD-1 knockout
Drug: PD-1 mAb — Patients will be treated with an identical course with a FDA approved monoclonal antibody against PD-1
  Other Names: Keytruda
  Arms: PD-1 mAb
Other: Sham control — Patient's T cell will treated ex vivo with modification and then infused back in a similar time course.
  Arms: Sham Control

SUMMARY:
The study is to assess the safety and efficacy of the anti-MUC1 CAR T cells and /or PD-1 knockout engineered T cells for patients with advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
This is a combined phase 1 and 2 clinical study. The study is to assess the safety and efficacy of the anti-MUC1 CAR T cells and /or PD-1 knockout engineered T cells for patients with advanced non-small cell lung cancer. The treatment outcomes will be compared.

ELIGIBILITY:
Inclusion Criteria:

* MUC1 is expressed in malignancy tissues by immuno-histochemical (IHC).
* Eastern cooperative oncology group (ECOG) performance status of 0-1 or karnofsky performance status (KPS) score is higher than 60.
* Patients have a life expectancy > 12 weeks.
* Adequate venous access for apheresis or venous sampling, and no other contraindications for leukapheresis.
* Negative pregnancy test for females of child-bearing potentials.
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements: White blood cell count (WBC) ≥ 2500c/ml, Platelets ≥ 50×10^9/L, Hb ≥ 9.0g/dL, lymphocyte (LY) ≥ 0.7×10^9/L, LY% ≥ 15%, Alb ≥ 2.8g/dL, serum lipase and amylase < 1.5×upper limit of normal, serum creatinine ≤ 2.5mg/dL, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5×upper limit of normal, serum total bilirubin ≤ 2.0mg/dL. These tests must be conducted within 7 days prior to registration.
* Signed informed consent form.

Exclusion Criteria:

* Number of T cells is less than 10% or the amplification of the T cells via artificial antigen presenting cell (aAPC) stimulation is less than 5 times.
* Patients with symptomatic central nervous system (CNS) involvement.
* Pregnant or nursing women.
* Known HIV infection.
* Serious illness or medical condition which would not permit the patient to be managed according to the protocol, including active uncontrolled infection, major cardiovascular, coagulation disorders, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive/restrictive pulmonary disease, or psychiatric or emotional disorders.
* History of severe immediate hypersensitivity to any of the agents including cyclophosphamide, fludarabine, or aldesleukin.
* Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary.
* Previously treatment with any gene therapy products.
* The existence of unstable or active ulcers or gastrointestinal bleeding. Patients with portal vein vascular invasion or extrahepatic, are excluded from this study.
* Patients with a history of organ transplantation or are waiting for organ transplantation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events and dose limiting toxicities as assessed by CTCAE v4.0 | approximately 6 months
  Safety and tolerability of dose of CART-cells and PD-1 Knockout T cells will be assessed using CTCAE v4.0.

SECONDARY OUTCOMES:
Response Rate | 6 months
  Will be assessed according to the revised RECIST guideline v1.1
Overall Survival - OS | Up to 24 months
  Measure the time from enrollment to death
Progression free survival - PFS | Up to 12 months
  Time from enrollment to date of first documented progression or date of death.
Median CAR-T cell persistence | 4 years
  Will be measured by quantitative RT-PCR

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - Professor Size Chen, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barr T, Ma S, Li Z, Yu J. Recent advances and remaining challenges in lung cancer therapy. Chin Med J (Engl). 2024 Mar 5;137(5):533-546. doi: 10.1097/CM9.0000000000002991. Epub 2024 Feb 7. PMID 38321811